CLINICAL TRIAL: NCT00252421
Title: The Effects of Organic Nitrates on Osteoporosis: Part 2
Brief Title: The Nitrate and Bone Study: Effects of Nitrates on Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Sophie Jamal, Associate Professor/Endocrinologist, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-169; ISRCTN 94484747
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Osteoporosis
Keywords: osteoporosis; bone mineral density; nitrates
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitroglycerin (Active Comparator): Nitroglycerin ointment 15 mg/day daily for 24 month
  Interventions: Drug: Nitroglycerin ointment 15 mg/day daily for 24 month
- Placebo (Placebo Comparator): Placebo ointment daily for 24 month
  Interventions: Drug: Placebo ointment daily for 24 month

INTERVENTIONS:
Drug: Nitroglycerin ointment 15 mg/day daily for 24 month — Nitroglycerin ointment 15 mg/day applied daily for 24 mth
  Arms: Nitroglycerin
Drug: Placebo ointment daily for 24 month — Placebo ointment applied daily for 24 mth
  Arms: Placebo

SUMMARY:
Osteoporosis or "thinning of the bones" affects in 1 in 4 Canadian women and 1 in 8 Canadian men. Moreover, while the rates of osteoporosis among Canadians are stabilizing, worldwide the number of people afflicted with osteoporosis continues to rise. The most serious complication of osteoporosis is a broken bone or fracture. Fractures due to osteoporosis can result in long hospital stays, dependence on others, and premature death. While there are several medications that prevent osteoporosis they all have side effects. For example, postmenopausal women who take hormone replacement therapy (HRT) are at increased risk of breast cancer and heart disease. In addition, drugs to prevent osteoporosis are expensive and not available worldwide. Therefore, it is essential that researchers continue to identify and test new medications for the prevention of osteoporosis.

The purpose of the research is to determine if nitrates, a group of drugs that are widely available, inexpensive, and commonly used to treat chest pain or angina, can prevent osteoporosis in women. If the researchers find that nitrates prevent osteoporosis, a widely available, inexpensive treatment for osteoporosis prevention that does not have any long term side effects would have been identified. This will improve the health of patients with osteoporosis worldwide.

DETAILED DESCRIPTION:
This proposal consists of two studies. The objective of the first study is to determine which of isosorbide mononitrate (ISMO) at 20 mg/day or nitroglycerin ointment (NTG) at 15 mg/day results in fewer headaches. The nitrate that is best tolerated will be used in a second study with one main objective: To determine if postmenopausal women with a T-score at the lumbar spine (L1 to L4) between 0 and -2.0 randomized to two years of treatment with intermittent nitrates have a greater increase in spine BMD as compared to women randomized to placebo.

We hypothesize that:

1. Women will report fewer headaches when they are randomized to intermittent NTG ointment at 15 mg/day compared to intermittent oral ISMO at 20 mg/day.
2. After two years, women randomized to intermittent nitrates will have a greater percent increase in lumbar spine BMD compared with women randomized to placebo.

To test these hypotheses we will execute 2 trials both of which include postmenopausal women, aged 50 and older, with BMD T scores at the lumbar spine between 0 and -2.0. We will exclude subjects with prior osteoporotic fractures or OP by BMD testing, subjects with current metabolic bone or cardiovascular disease, subjects taking treatments for OP, subjects with migraine headaches, and subjects with known hypersensitivity to nitrates. We will use computer generated randomization to allocate subjects to treatment assignments. To avoid bias the studies will be double-blind. The first study, which uses a crossover design, will recruit 22 subjects who will be randomly assigned to each of NTG ointment and ISMO for one week. In between treatments there will be a two week wash out period. Subjects will rate headaches on a daily basis using a visual analog scale and for each subject I will calculate the mean headache score over the 7 day treatment period for both treatments. We will then calculate the mean headache score (considering all subjects) for NTG and the mean headache score for ISMO. We will compare the mean headache scores for both treatments and the nitrate preparation that is best tolerated (lowest mean score) will be used in a second placebo controlled study (the main study) whose primary objective is to assess the effects of intermittent nitrates on spine BMD (L1 to L4) in 280 postmenopausal women. To limit differential drop out due to headaches among subjects randomized to nitrates, the main trial will follow a run-in phase during which all subjects will receive nitrates for one week. Only those subjects who do not have headaches resulting in discontinuation of the study medication during the nitrate run-in phase will enter the main study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50 and older
* Lumbar spine BMD (L1 to L4) T score between 0 and -2.0
* At least 3 years postmenopausal

Exclusion Criteria:

* Prior low trauma hip or vertebral fracture
* Total hip or femoral neck T score of <-2.0
* Bone disorders other than osteopenia (e.g., hyperparathyroidism or Paget's disease)
* Treatment within six months of study entry with androgen, calcitonin, estrogen, progesterone, fluoride in a tablet form, raloxifene, tamoxifen, etidronate, prednisone or an equivalent at 5 mg/d for 12 months or greater, lithium or anticonvulsants
* Alendronate or risedronate use for at least four weeks, within the last three years
* Current treatment with nitrates
* Systolic blood pressure of =<100 mm Hg or diastolic blood pressure >=100 mm Hg at the baseline screening examination
* Abnormal electrocardiogram (ECG) at the baseline screening examination
* history of myocardial infarction, angina, valvular or congenital heart disease
* Disabling conditions that may interfere with follow-up visits
* Inability to give informed consent
* Migraine headaches
* Hypersensitivity to nitrates

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2005-10; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pilot Study: Mean headache score associated with each of intermittent nitroglycerin ointment (NTG) and isosorbide mononitrate (ISMO) use | 6 months
Main Study: Change from baseline in bone mineral density (BMD) at the lumbar spine over 24 months | 48 months

SECONDARY OUTCOMES:
Change from baseline in total hip BMD; Change from baseline in bone formation and bone resorption markers; Adverse events and Bone microarchitecture: trabecular and cortical volumetric bone densities at the radius and tibia. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie A. Jamal, MD, PhD, Principal Investigator — Women's College Hospital, St. Michael's Hospital, University of Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Jamal SA, Cummings SR, Hawker GA. Isosorbide mononitrate increases bone formation and decreases bone resorption in postmenopausal women: a randomized trial. J Bone Miner Res. 2004 Sep;19(9):1512-7. doi: 10.1359/JBMR.040716. Epub 2004 Jul 26. PMID 15312252